CLINICAL TRIAL: NCT06570811
Title: Effect of Coenzyme Q10 (COQ10) on Chemotherapeutic Toxicity in Cancer Patients
Brief Title: Coenzyme Q10 and Chemotherapeutic Toxicity in Breast Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Damanhour University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COQ10 Breast Cancer Study
Record Dates: First submitted 2024-08-09; First posted 2024-08-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Chemotherapeutic Toxicity
MeSH Terms: conditions — Breast Neoplasms | interventions — coenzyme Q10; ubiquinol

STUDY DESIGN:
Intervention Model Description: This study is a parallel study
Masking Description: This is an open label study where Patients will be classified as follow:
  Control arm :20 Patients will receive 80 mg/m2 of paclitaxel chemotherapy weekly for 12 weeks after receiving 4 cycles of AC protocol (Adriamycin and cyclophosphamide)
  Treatment arm : 20 Patients will receive the same regimen as group1 in addition to 200 mg Coenzyme Q10 twice daily for 3 months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Comparator (Experimental): Placebo Group: 20 patients will receive 80 mg/m2 of paclitaxel chemotherapy weekly for 12 weeks after receiving 4 cycles of AC protocol (Adriamycin and cyclophosphamide)
  Interventions: Drug: Placebo
- Active Comparator (Experimental): Coenzyme Q10 Group : 20 patients will receive paclitaxel weekly for 12 weeks after receiving 4 cycles of AC protocol (Adriamycin and cyclophosphamide) in addition to oral 200 mg Coenzyme Q10 twice daily for 3 months.
  Interventions: Drug: Coenzyme Q10 200mg twice daily

INTERVENTIONS:
Drug: Placebo — Placebo tablets is supplied to breast cancer patients who receive 80 mg/ m2 paclitaxel (taxol®) chemotherapy.
  Arms: Placebo Comparator
Drug: Coenzyme Q10 200mg twice daily — 400 mg daily (200mg twice daily) of Coenzyme Q10 (an antioxidant that's in many foods, and it's made naturally in the investigator's bodies) is supplied to breast cancer patients who receive 80 mg/ m2 paclitaxel (taxol®) chemotherapy.
  Other Names: Coenzyme Q10 (Ubiquinol) -200mg ®
  Arms: Active Comparator

SUMMARY:
investigating the potential effect of Coenzyme Q10 in ameliorating and preventing the development of paclitaxel chemotherapeutic toxicity in breast cancer patients

DETAILED DESCRIPTION:
Fifty female patients with newly diagnosed breast cancer scheduled for weekly paclitaxel chemotherapy (80 mg/m2) will be randomized in a 1:1 ratio. The CoQ10 Group will receive Coenzyme Q10 supplementation (200 mg twice daily) for twelve weeks, while the Control Group will receive standard chemotherapy alone.

Safety monitoring for chemotherapy-related toxicities will be conducted using a multi-modal approach. Laboratory assessments, including complete blood counts (CBC) with differential, liver function, and renal function tests, will be obtained at baseline and prior to each weekly treatment cycle. Echocardiography will be performed at baseline and upon completion of the final cycle.

Hematological and non-hematological adverse events will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE), version 5.0. Non-hematological events (including fatigue, neuropathy, and gastrointestinal symptoms) will be captured via structured face-to-face interviews before each chemotherapy session and supplemented by a structured telephone follow-up three days after each session to reduce recall bias. Alopecia and nail changes will be monitored at baseline and at the end of the 12-week chemotherapy course.

ELIGIBILITY:
Inclusion Criteria:

1. women with newly diagnosed breast cancer r ≥18 years old.
2. Naive to chemotherapy.
3. Eastern Cooperative Oncology Group (ECOG) performance status from 0-2

Exclusion Criteria:

1. Advanced liver disease (defined as liver enzyme elevation >3-fold upper limit of normality, or cirrhosis); chronic kidney disease (CKD, defined as an estimated glomerular filtration rate (eGFR) <60 ml min-1 1.73 m-2).
2. Patients with a history of allergy to Coenzyme Q10 and similar compounds.
3. Concomitant use of opioids, anticonvulsants, tricyclic antidepressants, other neuropathic pain medication.
4. Pregnancy or breast feeding.
5. hereditary muscle disorders.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female breast cancer patients
Enrollment: 40 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events as Assessed by CTCAE v5.0 | 3 months
  The primary endpoint is Identtifying he number of participants experiencing chemotherapy-related toxicities including fatigue, sleep disturbance, peripheral neuropathy, nausea, vomiting, mucositis, anemia, febrile neutropenia, and pruritus. Grading is based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0.The grades as follow
  * Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  * Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate Instrumental activities of daily living (IADL)
  * Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL.
  * Grade 4 Life-threatening consequences; urgent intervention indicated.
  * Grade 5 Death

CONTACTS AND LOCATIONS:
Overall Officials: Amira B Kassem, PhD, Study Chair — Ass.professor in clinical pharmacy ,Faculty of pharmacy Damanhour university; Noha Ahmed El Bassiouny, PhD, Study Chair — Ass.professor in clinical pharmacy ,Faculty of pharmacy Damanhour university; Ahmed Ashour, PhD, Study Director — Lecturer in oncology , Faculty of mediciné Alexandria University; Yasser Abdelkader, Study Director — Head of oncology department, Damanhour Oncology Center; Gehad Hassoub, Bachelor, Principal Investigator — Teaching assistant in clinical pharmacy, faculty of pharmacy, Damanhour university
Locations (1):
- Damanhour Oncology Center, Damanhūr, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haroun EA, Mansour NO, Eltantawy A, Shams MEE. Effect of cilostazol on preventing paclitaxel-induced neuropathy in patients with breast cancer: A randomized controlled trial. Pharmacotherapy. 2023 Sep;43(9):872-882. doi: 10.1002/phar.2830. Epub 2023 Jun 12. PMID 37199288
- [Background] Bakry HM, Mansour NO, ElKhodary TR, Soliman MM. Efficacy of metformin in prevention of paclitaxel-induced peripheral neuropathy in breast cancer patients: a randomized controlled trial. Front Pharmacol. 2023 Jul 31;14:1181312. doi: 10.3389/fphar.2023.1181312. eCollection 2023. PMID 37583905
- [Background] Hernandez-Ojeda J, Cardona-Munoz EG, Roman-Pintos LM, Troyo-Sanroman R, Ortiz-Lazareno PC, Cardenas-Meza MA, Pascoe-Gonzalez S, Miranda-Diaz AG. The effect of ubiquinone in diabetic polyneuropathy: a randomized double-blind placebo-controlled study. J Diabetes Complications. 2012 Jul-Aug;26(4):352-8. doi: 10.1016/j.jdiacomp.2012.04.004. Epub 2012 May 16. PMID 22595020
- [Background] Khalefa HG, Shawki MA, Aboelhassan R, El Wakeel LM. Evaluation of the effect of N-acetylcysteine on the prevention and amelioration of paclitaxel-induced peripheral neuropathy in breast cancer patients: a randomized controlled study. Breast Cancer Res Treat. 2020 Aug;183(1):117-125. doi: 10.1007/s10549-020-05762-8. Epub 2020 Jun 29. PMID 32601973